CLINICAL TRIAL: NCT06218706
Title: A Randomized, Sham-Controlled Trial Investigating Low Intensity Focused Ultrasound as a Novel Treatment for Refractory Opioid Use Disorder
Brief Title: LIFU for Treatment for Refractory Opioid Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ali Rezai (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Ali Rezai, Director RNI, West Virginia University
Organization: West Virginia University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2312890071
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Randomization will occur after all inclusion criteria have been met at which time participants will be randomized 1:1 to either the Active or the Sham arm.
  After a participant completes the Week 12 post-LIFU study visit, that participant's treatment assignment is unblinded. Participants randomized to the Sham arm will be crossed over and receive Active LIFU after specified baseline procedures/assessments
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will occur after all inclusion criteria have been met at which time participants will be randomized 1:1 to either the Active or the Sham arm.This study will be performed in a double-blind manner, with participants as well as investigators and study staff involved with assessments unaware of treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- LIFU Treatment (Experimental)
  Interventions: Device: Low Intensity Focussed Ultrasound
- Sham treatment (Sham Comparator)
  Interventions: Device: Low Intensity Focussed Ultrasound

INTERVENTIONS:
Device: Low Intensity Focussed Ultrasound — The major objective of this study is to further test safety, tolerability, and feasibility of LIFU in this population as well as investigate the impact of LIFU on opioid and other substance use. The primary endpoint is 90 days (Post-LIFU Week 12) following Active/Sham LIFU. After the primary endpoint is reached, the blind will be broken and the group who received Sham LIFU will cross-over and receive Active LIFU

SUMMARY:
This is a randomized, double-blind, sham-controlled, partial crossover study investigating LIFU targeting the NAc and VC for participants with severe, treatment refractory OUD.

DETAILED DESCRIPTION:
The overall objective of this study is to assess the safety, tolerability, and feasibility of using Low Intensity Focused Ultrasound (LIFU) to treat opioid use disorder (OUD) as well as investigate the potential impact on substance use and risk factors associated with drug use recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Aged 22 - 60 years at time of enrollment.
* Fulfill current DSM-5 (American Psychiatric Association diagnostic and statistical manual of mental disorders, 5th ed, 2013) diagnostic criteria for severe OUD with at least a 2-year history.
* Women of reproductive potential must have negative pregnancy test and agree to use acceptable forms of contraception.

Exclusion Criteria:

* Unable to undergo MR-imaging because of non-MR compatible implants (e.g., pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent make-up or small metal fragments in the eye that welders and other metal workers may have), or if candidates are uncomfortable in small spaces (have claustrophobia) or cannot lie comfortably on their back for 2-3 hours.
* History of any clinically significant neurological disorder (e.g., brain surgery, tumors, uncontrolled epilepsy, or any others deemed clinically significant by the investigator).
* History of stroke or brain lesion in the targeted brain region (the NAc, ventral striatum, or VC).
* Implanted neurostimulators (e.g., vagus nerve stimulator, spinal cord stimulator, DBS).
* Documentation of clinically significant MRI abnormality indicative of a neurological condition or abnormality that may jeopardize the participant's safety, study conduct, or confound the participant's diagnostic assessments.
* More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp.
* Subject with chronic pulmonary disorders e.g. severe emphysema, pulmonary vasculitis, or other causes of reduced pulmonary vascular cross-sectional area.
* Subject with impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2
* Hepatic function laboratory values which are > 1.5 times the upper limit of normal unless deemed not clinically significant by a study investigator.
* Past or present diagnosis of schizophrenia or psychotic disorder.
* Subject unwilling to attempt abstinence from illicit substance use during the course of the study.
* Unable to speak, read and understand English.
* Subject is considered to be a poor surgical or study candidate, which may include, but is not limited to the following: any medical, social, or psychological problem that could complicate the required procedures and evaluations of the study in the judgment of the investigator.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Treatment Emergent Adverse Events | Post-ExAblate Procedure through 90 day Follow-Up
  Safety will be assessed by recording all adverse events that are treatment related. Each Adverse Event will be documented for patterns of occurrence.
Changes in Opioid Use | Post-ExAblate Procedure through 90 day Follow-Up
  Changes in opioid use will be measured using quantitative urine toxicology via liquid chromatography/mass spectrometry (LC/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rezai, Principal Investigator — Executive Director WVU Rockefeller Neuroscience Institute
Locations (1):
- WVU Rockefeller Neuroscience Institute, Morgantown, West Virginia, United States